CLINICAL TRIAL: NCT03129685
Title: Short-term Outcome of Ipsilateral Liver Lobe Devascularization of the Large Hepatocellular Carcinoma
Brief Title: Ipsilateral Liver Lobe Devascularization of the Large Hepatocellular Carcinoma
Acronym: NRU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The National Ribat University (Other)
Responsible Party: Principal Investigator, Osama Mohamed Elsanousi, Associate Professor of Surgery, The National Ribat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS-001-17
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Devascularization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Prospective and non-randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Devascularization (Experimental): Patients undergoing ipsilateral hepatic artery ligation with extrahepatic collaterals division (HALED)
  Interventions: Procedure: HALED

INTERVENTIONS:
Procedure: HALED — This is attained via a laparotomy involves isolation of the arterial blood supply of the tumor-containing liver lobe (the ipsilateral hepatic artery as well as the extrahepatic arterial collaterals) while preserving the feeding veins.

SUMMARY:
Assessment of short-term outcomes of ipsilateral lobe arterial devascularization of the large hepatocellular carcinoma: single center non-randomized trial.

DETAILED DESCRIPTION:
Assessment of the 30-day mortality and major complications as well as the tumor size changes of the patients undergoing ipsilateral lobe arterial devascularization of the large hepatocellular carcinoma. This is a prospective non randomized trial carried out at the Ribat University Hospital between April 2017 to March 2018.

ELIGIBILITY:
Inclusion Criteria:

* Review and sign informed consent;
* Between 15 and 80 years of age at time of trial enrollment;
* Documented pathological and/or radiological diagnosis of hepatocellular carcinoma;
* Radiologically documented tumor size of > 5 centimeters;
* Radiologically documented liver cirrhosis.

Exclusion Criteria:

* American Anesthesia Association (ASA) Class IV or V and/or any contraindications to general anesthesia;
* Uncontrollable ascites;
* Deep persistent jaundice;
* Hepatic encephalopathy;
* Coagulopathy;
* Severe thrombocytopenia;
* Unable or unwilling to attend follow up visits and examinations;
* Other associated surgical procedure;

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-11-19 (Estimated); Study Completion 2018-12-19 (Estimated)

PRIMARY OUTCOMES:
Short term mortality rate | 30 day
  Percentage of patients' postoperative deaths

SECONDARY OUTCOMES:
Short term major complications' rate | 30 days
  Incidence of Clavien/Dindo grade 3 or more postoperative complications
Tumor response rate according to mRECIST criteria. | 30 days
  Estimation of the residual percentage of viable tumor following the devascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Elsanousi, MD, Principal Investigator — Faculty of Medicine. The National Ribat University
Locations (1):
- Ribat University Hospital, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From June 2018 - December 2018
Access Criteria: Free

REFERENCES:
- [Derived] Elsanousi OM, Mohamed MA, Salim FH, Adam EA. Selective devascularization treatment for large hepatocellular carcinoma: Stage 2A IDEAL prospective case series. Int J Surg. 2019 Aug;68:134-141. doi: 10.1016/j.ijsu.2019.06.014. Epub 2019 Jun 29. PMID 31265917